CLINICAL TRIAL: NCT02227199
Title: A Phase I/II Trial of Brentuximab Vedotin (BV), Ifosfamide (I), Carboplatin (C), and Etoposide (E) for Patients With Relapsed or Refractory Hodgkin Lymphoma (BV-ICE)
Brief Title: Brentuximab Vedotin, Ifosfamide, Carboplatin, and Etoposide in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma
Acronym: BV-ICE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Seagen Inc. (Industry)
Responsible Party: Principal Investigator, Ajay Gopal, Professor, Department of Medicine, Division of Oncology, University of Washington
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9111; NCI-2014-01782 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9111 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1714038 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Carboplatin; Etoposide; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) (Experimental): Patients receive brentuximab vedotin 1.2mg/kgIV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Interventions: Drug: Brentuximab Vedotin; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis
- Phase I: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) (Experimental): Patients receive brentuximab vedotin 1.5mg/kgIV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Interventions: Drug: Brentuximab Vedotin; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis
- Phase II: Dose Expansion (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) (Experimental): Patients receive brentuximab vedotin 1.5mg/kgIV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Interventions: Drug: Brentuximab Vedotin; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of brentuximab vedotin that can be combined with ifosfamide, carboplatin, and etoposide in treating patients with Hodgkin lymphoma that has come back (relapsed) or is not responding to treatment (refractory). Monoclonal antibody-drug conjugates, such as brentuximab vedotin, can block cancer growth in different ways by targeting certain cells. Chemotherapy drugs, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving brentuximab vedotin together with an ifosfamide, carboplatin, and etoposide chemotherapy regimen may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine maximally tolerated dose of brentuximab vedotin that can be combined with ifosfamide, carboplatin and etoposide chemotherapy in patients with relapsed or refractory Hodgkin lymphoma.

II. To gain a preliminary assessment of the efficacy of the above regimen.

SECONDARY OBJECTIVES:

I. To determine the safety and toxicity of the above regimen.

II. To determine the ability to proceed to peripheral blood stem cell collection following the above regimen (the impact of above regimen on stem cell reserve).

III. To assess the impact of this regimen on biomarkers from the microenvironment in Hodgkin lymphoma tumors.

OUTLINE: This is a phase I, dose-escalation study of brentuximab vedotin followed by a phase II study.

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative high-dose therapy (HDT) and autologous stem cell transplantation (ASCT) may undergo peripheral blood stem cell (PBSC) mobilization following the 2nd course of study therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have primary refractory or first relapse of cluster of differentiation 30 (CD30)+ Hodgkin lymphoma
* Patients must have measurable disease defined as lesions that can be accurately measured in two dimensions by computed tomography (CT), magnetic resonance imaging (MRI), medical photograph (skin or oral lesion), plain x-ray, or other conventional technique and a greatest transverse diameter of 1 cm or greater; or palpable lesions with both diameters >= 2 cm; further, at least 1 of these lesions must be positive by positron emission tomography (PET) scan (i.e., Deauville score of 4 or more); Note: CT scans remain the standard for evaluation of nodal disease
* Patients must have a CT of chest, abdomen, and pelvis with PET within 28 days of enrollment; patients with evidence of lymphadenopathy in the neck must have a dedicated CT of neck
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (performance status of 2 will be allowed if poor performance status is thought to be directly secondary to patient's Hodgkin lymphoma [HL])
* Absolute neutrophil count (ANC) >= 1,500/uL, performed within 28 days prior to registration
* Platelets >= 100,000/uL (without transfusion or growth factor support), performed within 28 days prior to registration
* Serum creatinine < 1.5 mg/dl or creatinine clearance (CrCl) > 60 mL/min, performed within 28 days prior to registration
* Total bilirubin < 2 times upper limit of normal (unless due to Gilbert's syndrome), performed within 28 days prior to registration
* Aspartate aminotransferase (AST) < 2.5 times upper limit of normal, performed within 28 days prior to registration
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Patients must be anticipated to complete 2 cycles of chemotherapy

Exclusion Criteria:

* Patients known to be positive for human immunodeficiency virus (HIV)
* Pregnant or nursing women; men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, breast or cervical cancer in situ, or other cancer from which the patient has been disease-free for 5 years or greater, unless approved by the protocol chair or co-chair
* Patients with known allergy, intolerance, or resistance (i.e., remission duration less than 6 months or lack of response) to ifosfamide, carboplatin, or etoposide
* Patients with evidence of active central nervous system lymphoma
* Patients with prior receipt of brentuximab vedotin
* Patients with peripheral neuropathy of > grade 1
* Patients who have other medical conditions that would contraindicate treatment with aggressive chemotherapy (including active infection, uncontrolled hypertension, congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or uncontrolled arrhythmia); if the patient's cardiac history is questionable, a measurement of left ventricular ejection fraction should be obtained within 42 days prior to registration; patients with left ventricular ejection fraction < 50% are not eligible
* Prior failed (< 5 x 10^6 CD34/kg) peripheral blood stem cell (PBSC) collection
* Patients who had pelvic radiation within 12 months
* Previous chemotherapy/immunotherapy within 3 weeks before study entry
* Concurrent use of other anti-cancer agents or experimental treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2025-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Lynch RC, Cassaday RD, Smith SD, Fromm JR, Cowan AJ, Warren EH, Shadman MS, Shustov A, Till BG, Ujjani CS, Libby EN 3rd, Philip M, Coye H, Martino CN, Bhark SL, Morris K, Rasmussen H, Behnia S, Voutsinas J, Gopal AK. Dose-dense brentuximab vedotin plus ifosfamide, carboplatin, and etoposide for second-line treatment of relapsed or refractory classical Hodgkin lymphoma: a single centre, phase 1/2 study. Lancet Haematol. 2021 Aug;8(8):e562-e571. doi: 10.1016/S2352-3026(21)00170-8. PMID 34329577

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide): Patients receive brentuximab Vedotin 1.2mg/kg IV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Brentuximab Vedotin: Given IV
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide); Phase 2: Dose Expansion (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide): Patients receive brentuximab Vedotin 1.5mg/kg IV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Brentuximab Vedotin: Given IV
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) | Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) | Phase 2: Dose Expansion (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide)
Started | 3 | 3 | 39
Completed | 3 | 3 | 35
Not Completed | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Escalation, Dose Level 1 (Brentuximab 1.2mg/kg, Ifosfamide, Carboplatin, Etoposide) | Phase I: Dose Escalation, Dose Level 2 (Brentuximab 1.5mg/kg, Ifosfamide, Carboplatin, Etoposide) | Phase II: Dose Expansion (Brentuximab 1.5mg/kg, Ifosfamide, Carboplatin, Etoposide) | Total
Number analyzed (Participants) | 3 | 3 | 39 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 39 | 45
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 27 | 29
  Male | 1 | 3 | 12 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 3 | 3 | 35 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 3 | 32 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 39 | 45

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Brentuximab Vedotin That Can be Combined With Ifosfamide, Carboplatin, and Etoposide Chemotherapy
Description: Will be defined as the dose at which =< 1 of 6 patients experience a dose-limiting toxicity. Dose-limiting toxicity will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 28 days following the second course of chemotherapy, approximately 70 days
Measure: Number; unit: mg/kg
Groups:
- Treatment (brentuximab, ifosfamide, carboplatin, etoposide): Patients receive brentuximab vedotin IV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Brentuximab Vedotin: Given IV
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Treatment (brentuximab, ifosfamide, carboplatin, etoposide)
Number analyzed (Participants) | 6
mg/kg | 1.5

2. Primary Outcome: Percentage of Patients That Achieve a Complete Remission Following Study Treatment
Time Frame: 3 weeks following the completion of chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide); Phase II: Dose Expansion (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide): Patients receive brentuximab Vedotin 1.5mg/kg IV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Brentuximab Vedotin: Given IV
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) | Phase I: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) | Phase II: Dose Expansion (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide)
Number analyzed (Participants) | 3 | 3 | 39
Participants | 3 | 3 | 26

3. Secondary Outcome: 2 Year Overall Survival
Time Frame: Up to 2 years from initiation of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) | Phase I: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) | Phase II: Dose Expansion (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide)
Number analyzed (Participants) | 3 | 3 | 39
Participants | 3 | 3 | 37

4. Secondary Outcome: 2 Year Progression-free Survival
Time Frame: Up to 2 years from initiation of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) | Phase I: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) | Phase II: Dose Expansion (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide)
Number analyzed (Participants) | 3 | 3 | 39
Participants | 2 | 3 | 33

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting after the first dose of study treatment and collected through 30 days after the last dose of study drug, or until the patient receives an alternative anti-cancer therapy, whichever date comes first, approximately 60 days.
Groups:
- Phase 1: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide): Patients receive brentuximab vedotin 1.2mg/kg IV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Brentuximab Vedotin: Given IV
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Phase 1: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide): Patients receive brentuximab vedotin 1.5mg/kg IV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
  Brentuximab Vedotin: Given IV
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Phase 2: Dose Expansion, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide): Patients receive brentuximab vedotin 1.5mg/kg IV over 30 minutes on days 1 and 8; ifosfamide IV over 24 hours and carboplatin IV over 1 hour on day 2; and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients planning to go on to consolidative HDT and ASCT may undergo PBSC mobilization following the 2nd course of study therapy at the discretion of the treating physician.
Arm/Group | Phase 1: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) | Phase 1: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) | Phase 2: Dose Expansion, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 2/39
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 11/39
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) (N=3) | Phase 1: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) (N=3) | Phase 2: Dose Expansion, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) (N=39)
Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Elevated Lactate (Investigations) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Neutropenic Fever (General disorders) | 0 (0) | 0 (0) | 3 (3)
Septic Shock (Infections and infestations) | NA | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Sweet Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythematous Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation, Dose Level 1 (brentuximab 1.2mg/kg, ifosfamide, carboplatin, etoposide) (N=3) | Phase 1: Dose Escalation, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) (N=3) | Phase 2: Dose Expansion, Dose Level 2 (brentuximab 1.5mg/kg, ifosfamide, carboplatin, etoposide) (N=39)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 11 (13)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 12 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 19 (19)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 8 (10)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 10 (17)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 6 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (4) | 18 (19)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 10 (15)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 18 (23)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 29 (40)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 6 (7)
Platelet Count Decreased (Investigations) | 2 (3) | 1 (3) | 5 (8)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 12 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 6 (7)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (5) | 1 (1) | 15 (18)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 6 (7)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 4 (5)
Fatigue (General disorders) | 2 (4) | 3 (3) | 16 (19)
Fever (General disorders) | 1 (1) | 2 (2) | 4 (6)
Hiccups (General disorders) | 0 (0) | 0 (0) | 3 (3)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (8)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 11 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6)
Night Sweats (General disorders) | 0 (0) | 0 (0) | 5 (5)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 12 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (4)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 2 (4) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (5)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 7 (8)
Edema Limbs (General disorders) | 0 (0) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (3) | 1 (1) | 10 (12)
Neutrophil Count Decreased (Investigations) | 1 (1) | 1 (2) | 1 (1)
Pain at Hickman Site (General disorders) | 2 (2) | 1 (1) | 4 (4)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Flushing (General disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT02227199/Prot_SAP_000.pdf